CLINICAL TRIAL: NCT01587612
Title: Study of Quantification of Hyperpronation
Status: Completed | Type: Observational
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: ON-02-005-OSi
Record Dates: First submitted 2011-01-05; First posted 2012-04-30 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Foot Pain Chronic
Keywords: Pain; Foot
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
Hyperpronation is af frequent cause of excessive load in foot and crus. Pain and limited functional ability cause problems with work-related activities, sport activities and leisure activities.

There are only few studies of the frequency of pain related to hyperpronation in foot and the effect of exercises. Medics and physiotherapists need sufficient evidence-based knowledge to treat these patients correctly.

Therefore, the investigators want to study the effect of exercises and inner soles for treatment of patients with chronic pain and hyperpronation of foot.

ELIGIBILITY:
Inclusion Criteria:

* Hyperpronation of foot
* Consent of information

Exclusion Criteria:

* Normal gait
* Lack of consent of information
* Unable to speak and read Danish

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hyperpronation of foot
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2003-08; Primary Completion 2003-12 (Actual); Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mogens B Laursen, MD, Principal Investigator — Northern Orthopaedic Division
Locations (1):
- Northern Orthopaedic Division, Klinik Aalborg, Aalborg, Northern Jutland, Denmark